CLINICAL TRIAL: NCT03295968
Title: The Role of IL-6 in Exercise-Induced Anorexia in Normal-weight Boys
Brief Title: IL-6 in Exercise-Induced Anorexia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, G. Harvey Anderson, Professor, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: REB32277
Record Dates: First submitted 2017-09-22; First posted 2017-09-28 (Actual); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Appetitive Behavior; Pediatric Obesity
MeSH Terms: conditions — Appetitive Behavior; Pediatric Obesity | interventions — Ibuprofen

STUDY DESIGN:
Intervention Model Description: Fifteen normal-weight boys (aged 13-18y) were randomly assigned in a crossover design to four sessions: 1) Water + Rest; 2) Rest + ibuprofen; 3) Water + high intensity exercise; 4) high intensity exercise + ibuprofen. High intensity exercise consisted of three 10min bouts of high intensity exercise at 75% VO2peak at 60-70RPM with 1:30min active rest interposed. IBU was given in a 300mg liquid solution. EI, visual analog scale ratings and plasma biomarkers of appetite, inflammation, stress and glucose control were measured.
Who Masked: Participant
Masking Description: Water control and ibuprofen solution contained 0.8 g of Sucralose (Heartland Food Products Group, Amsterdam, HP, Netherlands) and 1.2 g of orange flavored Kool-Aid (Kraft Foods, Northfield, IL, United States) to mask the taste of the Motrin solution. To match sweetness and calorie content of the ibuprofen Motrin drink, the water control also contained 6 mL high fructose corn syrup (ACH Food Companies, Mississauga, ON, Canada).
Oversight: Data Monitoring Committee: No

ARMS (4):
- Water and Rest (No Intervention)
- Water and High Intensity Exercise (Experimental)
  Interventions: Other: High Intensity Exercise/Ibuprofen
- Ibuprofen and Rest (Experimental)
  Interventions: Other: High Intensity Exercise/Ibuprofen
- Ibuprofen and High Intensity Exercise (Experimental)
  Interventions: Other: High Intensity Exercise/Ibuprofen

INTERVENTIONS:
Other: High Intensity Exercise/Ibuprofen — HIEX, with and without the inflammation inhibitor, ibuprofen, on plasma levels of IL-6 and other selective biomarkers of inflammation and appetite on food intake and subjective ratings of appetite in normal-weight boys.
  Arms: Ibuprofen and High Intensity Exercise; Ibuprofen and Rest; Water and High Intensity Exercise

SUMMARY:
This study investigates the effect of high intensity exercise, with and without the inflammation inhibitor, ibuprofen, on plasma levels of IL-6 and other selective biomarkers of inflammation and appetite on food intake and subjective ratings of appetite in normal-weight boys.

ELIGIBILITY:
Inclusion Criteria:

* 13-18 yrs, healthy, male

Exclusion Criteria:

* female, heamatophobia, following a diete, diagnosed with diabetes or other metabolic diseases, scoring ≥11 on an Eating Habit Questionnaire

Ages: 13 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Fifteen normal-weight (BMI for age percentile: 15th-85th) boys aged 13-18yrs completed the study. Sample size was determined through previous studies in our lab. A telephone questionnaire was employed to determine eligibility for this study. Boys who answered "yes" to one of the questions of the physical activity readiness questionnaire, displayed a form of heamatophobia, dieters, have been diagnosed with diabetes or other metabolic diseases, and those scoring ≥11 on an Eating Habit Questionnaire were excluded from the study.
Enrollment: 15 (Actual)
Dates: Start 2016-03; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Food Intake | 100-120 min
  Participants were provided with ad libitum lunch meal, consisting of rice (Uncle Ben's, Bolton, ON, Canada), beef meatballs (President's Choice, Brampton, ON, Canada) and tomato sauce (Ragu, Mount Prospect, IL, USA) at 100 - 120 min. The meatballs were cut into small and uniform pieces and were mixed homogeneously with the other ingredients in a bowl. One bowl was a 479.5 g portion which represented 827.5 kcal, 30.8 g fat, 104.8 g carbohydrate and 30.2 g protein based on the weight consumed and the compositional information provided by the manufacturers. Two portions we served in 10 min intervals and FI from the pizza meal was calculated based on the weight consumed during the lunch. Participants were instructed to eat until comfortably and stay seated during the duration of the meal.
Visual Analog Scale Appetite Scores | 0-120min
  Visual Analog Scales were employed to assess subjective appetite based on the following questionnaires: Determination to Eat, Hunger, Fullness and Prospective Food Consumption.
Appetite Biomarkers | 0-120min
  Active Ghrelin, Blood Glucose, Insulin, Peptide-YY and Glucagon-like peptide-1 were determined as appetite biomarkers.
Inflammatory and Stress Biomarkers | 0-120min
  Interleukin-6, Tumor necrosis factor alpha and cortisol were determined as appetite biomarkers.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available to other researchers.Participant's identities will be kept confidential. Records will be kept in a locked filing cabinet in the Fitzgerald building at 150 College Street, room 437. Access will be restricted to those directly involved with the project, such as the investigator and the co-investigators. Following recruitment and attainment of informed consent, participants will be given an ID # which will be used on all forms and data analysis. Informed consent forms will be kept in a locked cabinet in a locked office, contain participant names. Research records will be identified by initials, ID number, test and date. Results identified by date and ID number will only be entered on password-protected personal computers kept in locked laboratories or offices at the University of Toronto. Any electronic data will be held on encrypted computers and USB sticks for the same period of time.

REFERENCES:
- [Background] Almada C, Cataldo LR, Smalley SV, Diaz E, Serrano A, Hodgson MI, Santos JL. Plasma levels of interleukin-6 and interleukin-18 after an acute physical exercise: relation with post-exercise energy intake in twins. J Physiol Biochem. 2013 Mar;69(1):85-95. doi: 10.1007/s13105-012-0191-x. Epub 2012 Jul 19. PMID 22810957
- [Background] Anderson GH, Hunschede S, Akilen R, Kubant R. Physiology of Food Intake Control in Children. Adv Nutr. 2016 Jan 15;7(1):232S-240S. doi: 10.3945/an.115.009357. Print 2016 Jan. PMID 26773031
- [Background] Banks WA. Anorectic effects of circulating cytokines: role of the vascular blood-brain barrier. Nutrition. 2001 May;17(5):434-7. doi: 10.1016/s0899-9007(01)00507-x. PMID 11377145
- [Background] Banks WA, Gertler A, Solomon G, Niv-Spector L, Shpilman M, Yi X, Batrakova E, Vinogradov S, Kabanov AV. Principles of strategic drug delivery to the brain (SDDB): development of anorectic and orexigenic analogs of leptin. Physiol Behav. 2011 Nov 30;105(1):145-9. doi: 10.1016/j.physbeh.2011.05.024. Epub 2011 Jun 6. PMID 21669216
- [Background] Blundell JE, Gibbons C, Caudwell P, Finlayson G, Hopkins M. Appetite control and energy balance: impact of exercise. Obes Rev. 2015 Feb;16 Suppl 1:67-76. doi: 10.1111/obr.12257. PMID 25614205
- [Background] Blundell JE, King NA. Exercise, appetite control, and energy balance. Nutrition. 2000 Jul-Aug;16(7-8):519-22. doi: 10.1016/s0899-9007(00)00250-1. No abstract available. PMID 10906542